CLINICAL TRIAL: NCT02891096
Title: Inspiratory Muscle Strength and Respiratory Complications After Spinal Cord Injury: a Multicenter, Prospective Cohort Study
Brief Title: Inspiratory Strength and Respiratory Complications After SCI Injury
Acronym: RESCOM
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Balgrist University Hospital (Other); Rehab Basel (Other); Clinique Romande de Readaptation (Network); Rehabilitation Clinic Tobelbad, Austria (Unknown); Rehabilitation Center Haering, Austria (Unknown); Austin Hospital, Melbourne Australia (Other); Erasmus Medical Center (Other); Heliomare Rehabilitation, Wijk aan Zee, The Netherlands (Unknown); BG Unfallklinik Murnau (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-14
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injuries; Pneumonia
Keywords: respiratory complications; respiratory muscle strength; discriminator
MeSH Terms: conditions — Spinal Cord Injuries; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: inspiratory muscle strength — Measurements:
  * in- and expiratory muscle strength (5min)
  * lung function (FVC, FEV1, PEF, PCF) (10 min)
  Questionnaires:
  * ISCoS core data-set
  * ISCoS pulmonary function data sets
  * ISCoS quality of life questionnaire
  * questionnaire on individual respiratory muscle training, regular physical exercise and therapies
  * individual medication/vaccination and other medical complications will be assessed from patient's medical records
  All measurements will be performed at each of the 4 measurement time-points (up to 4 times during inpatient rehabilitation) and last about 40 min per patient and measurement time-point in total (time with patient).

SUMMARY:
The investigators conducting this study to investigate the relation between the respiratory muscle strength and respiratory complications. To understand more about respiratory complications the influence of different factors (such as in- and expiratory muscle strength, lung function parameters, physical activity, smoking, medications,…) on respiratory complications (such as pneumonia) will be investigated.

DETAILED DESCRIPTION:
Background:

A spinal cord injury (SCI) often leads to paralysis of respiratory muscles (1), which causes a decrease in inspiratory volume and consequently limits the pre-cough volumes needed to produce an effective cough (2). The ability to cough is essential for airway clearance (3). With reduced cough capacity, the risk for pneumonia is increased (1). Pneumonia is still among the leading causes of death in the SCI population (4, 5). In acute SCI, up to 80% of patients are affected by respiratory complications (6) and in 51 % of these cases pneumonia occurs (7), corresponding to a cumulative pneumonia incidence rate of about 40%. Unfortunately, predictors of pneumonia in SCI are still poorly understood (6).

To the investigators knowledge, there are three studies on predictors of pneumonia in the SCI population (8, 9).

Two of these studies concentrated on factors of injury and shock severity (9) or identified the level and completeness of injury as the fundamental clinical entity predicting pulmonary complications (8).

However, both studies did not investigate potentially modifiable factors. The third study focused on potentially modifiable factors, such as lung function but did not cover respiratory muscle strength and did not define the inclusion of respiratory complications precisely (10). Therefore, to facilitate future evidence-based strategies to reduce the pneumonia risk in acute SCI, prevention targeted studies that aim to identify modifiable risk factors for pneumonia are urgently needed.

The current research proposal is targeted at specific parameters of respiratory function that are conceivably determinants of pneumonia risk as well as modifiable by respiratory muscle training (11,12). In a recent study (EKNZ 2014-293; accepted for Publication in Respiratory Care) the investigators evaluated various respiratory function parameters and identified inspiratory muscle strength as a reliable discriminator between individuals with and those without pneumonia.

Although the investigators identified inspiratory muscle strength as best parameter of respiratory function to discover individuals with SCI at risk for pneumonia, these data are based on a retrospective singlecenter data analysis without any detailed information on the type, time-point and severity of pneumonia. Also data on mortality due to pneumonia and other personal parameters that may influence the risk for pneumonia as well (e.g. smoking, exercise, mechanical ventilation dependency etc.) are missing in this analysis.

Objective:

The main objective of this study is to evaluate 'cut-off levels' of inspiratory muscle strength as predictor for pneumonia in individuals with SCI (diagnostic accuracy). Additionally, to evaluate lifestyle and treatment parameters as well as personal- and lesion characteristics as further potential determinants of pneumonia as well as the impact of pneumonia on quality of life and mortality.

Determination of sample size:

Regarding the in- and exclusion criteria, the investigators made a calculation of a realistic number of subjects who can be recruited for this study per year and center, based on the number of patients admitted to the corresponding center during the last years. Overall, the investigators will be able to recruit about 250 patients per year for this study.

With an anticipated number of 625 subjects over a 2.5 years recruitment period, the investigators may detect about 250 cases of pneumonia (under the assumption of a 40% incidence rate (6,7). Moreover, taking the diagnostic accuracy (i.e., area under the curve (AUC of 0.86 from a retrospective study as reference, the envisioned sample size of at least 250 cases per diagnostic group should allow for detecting a diagnostically and clinically relevant effect (i.e., change in AUC) of 0.07 to 0.05 with 95% confidence level and 80% power (18).

Criteria for withdrawal:

Reasons for which a participant needs to discontinue from the project:

* withdrawal of informed consent
* non-compliance
* medical complications which do not allow measurements of this study
* death

In case of drop-out, the already recorded data will be used for further analyses. All data of drop-out patients will be anonymized after analysis.

The investigators will report all reasons for withdrawal of the participants and compare the reasons qualitatively.

The study will not be stopped in case of futility, unless CTU Nottwil during the course of safety monitoring advices otherwise. In this case, CTU Nottwil will discuss potential stopping for futility with the study investigators group.

The final decision to terminate the study is taken by the Principal Investigator of the study RESCOM.

Risk-Benefit:

Patients have to perform a maximum of 4 measurement sessions (dependent on the time of rehabilitation) with 15 min of measurements each. Therefore the time needed for this study will not negatively influence rehabilitation of included patients. Respiratory muscle strength measurements and cough capacity measurements are non-invasive and also part of clinical routine. Safety of these measurements is very high and to the best of our knowledge the investigators are not aware of any adverse Events due to such measurements.

Potential benefit of project result:

Increased knowledge on determinants and effects of pneumonia will help adapt rehabilitative strategies/therapy to prevent patients from pneumonia and thereby also increase quality of life of the patients and life expectancy.

Methods of minimising bias:

Throughout the study, the coding of the participants will be conducted by the study nurses of each site in order to keep the data management and the biostatistician blind against the study condition as long as the data base is open.

The coding list remains with the study nurses of each site for the whole duration of the study. Thus, coding will be conducted without any influence of the principal investigator or raters.

The study investigators will strive for complete separation of the individuals involved in the steps before enrolment from those involved in the data management and analysis.

Assessments of primary and secondary outcomes will be conducted by a study nurse without any influence on data analysis. All study nurses will go through a profound assessment training program.

A study nurse will enter data into the secuTrial® data management system so that the biostatistician can analyze the data without having access to information about the origin, or names of participants.

Assessment of safety and reporting:

An annual safety report will be submitted once a year to the local Ethics Committee via local Investigator.

For multi-center studies the annual safety report contains information from all sites including information from sites outside of Switzerland. The Sponsor-Investigator prepares it, and then submits it to the participating Investigators. The participating Investigators submit it to the local committees.

Statistical considerations:

To evaluate the diagnostic accuracy of markers of lung function (particularly MIP) for predicting or excluding clinical pneumonia the investigators will use contemporary receiver operating characteristic (ROC) analyses techniques that allow for adjusting of covariate effects. Univariable and multivariable regression modelling will be used to evaluate the primary outcome and secondary outcomes. Multivariable modelling as compared univariable modelling will principally allow the investigators to investigate relative contribution of different predictors (or risk factors) to the outcome of interest, while controlling for potential confounding by other factors. Multivariable models may further be used to examine effect modification (interaction) as well as mediation.

Missing data:

Regression analyses of the primary outcome and secondary outcomes may suffer from missing data, which may cause bias and loss of information in analyses that are restricted to study participants with complete data ("complete-case analyses"). To appropriately account for missing data in advanced regression analyses the investigators will use multiple imputation techniques as well as an iterative imputation method (missForest) based on a random forest. Due to the relatively high anticipated sample size, the analysis will be split up into specific sub-Groups (e.g. completeness of lesion, para-/tetraplegia, type of pneumonia). For mortality flexible parametric modeling of survival data) and other secondary outcome analyses will be performed.

Data handling and record keeping/ archiving The secuTrìal data management system (iAS, Berlin, Germany), a web-based data capture and management system, will be used. The system is hosted on a server of the Swiss Paraplegic Centre.

The project set-up and eCRFs will be tested by the Data Manager of the Swiss Paraplegic Center, Clinical Trial Unit prior to the release into the productive environment using a custom testing protocol.

Every staff member is authorized for any CRF entry and by initials noted on the CRF the investigator can be subsequently identified. The data on the CRF will later be entered in the secuTrial database (iAS, Berlin, Germany).

One person will enter the data from the CRF paper form into the secuTrial database. A second person will control the correctness of the data in the secuTrial and the principal investigator will finally release the data for archival storage.

The Clinical Trial Unit will only give access to 2 people per center: Person A will get access for data entering and controlling and the local investigator (Person B) for data release.

Plausibility rules will be established in the data capture system to promote data quality. Furthermore, data will be reviewed and verified prior to data entry completion.

Encrypted data will be exported from the data management system for analysis in statistic software.

Data protection:

Project data will be handled with uttermost discretion and only be accessible to authorized personnel.

Direct access to source documents will be permitted for purposes of monitoring, audits or inspections.

The data management system allows to define roles for data entry, verification, validation and management. An audit trail documents all entries and changes made in the system and by whom.

Personal data of participating subjects which allow to identify an individual, will not be stored on a server or personal computer, nor will any names of subjects be transmitted to the main study center in Nottwil. These data will be printed on paper and stored in a locked data storage room with limited access in each participating center. An anonymous identification number will allow to connect the data entered in the system, but only by each center for their own subjects. Only anonymous data will be stored in the electronic data capture and management system. Encrypted data will be exported from the data management system for analysis in statistic software.

For data verification purposes, authorized representatives of a competent authority (e.g. an ethics committee) may require direct access to parts of the medical records relevant to the project, including participants' medical history.

ELIGIBILITY:
Inclusion Criteria:

* Initial rehabilitation after SCI
* men and women
* aqe over or equal 18 years
* AIS A, B, C or D lesion
* lesion level C1-T12

Exclusion Criteria:

* Neurologic diseases (e.g. MS, ALS)
* 24h mechanical ventilation dependency
* mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with spinal cord injury during primary inpatient rehabilitation in a specialized center.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Mueller, PhD, Principal Investigator — Swiss Paraplegic Centre Nottwil, Clinical Trial Unit
Locations (1):
- Swiss Paraplegic Centre Nottwil, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
In general, only the study investigators have access to the full study dataset in order to ensure that the overall results are not disclosed by an individual study site prior to the main publication. Site investigators are allowed to access the full dataset if a formal request describing their plans is approved by the study investigators.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 1.1.2025 until 31.12.2029
Access Criteria: official collaborating center ot this study or personnal request of data at the study center (PI) based on a clear hypothesis, protocol and analysis plan.

REFERENCES:
- [Background] Lanig IS, Peterson WP. The respiratory system in spinal cord injury. Phys Med Rehabil Clin N Am. 2000 Feb;11(1):29-43, vii. PMID 10680156
- [Background] Kang SW, Bach JR. Maximum insufflation capacity: vital capacity and cough flows in neuromuscular disease. Am J Phys Med Rehabil. 2000 May-Jun;79(3):222-7. doi: 10.1097/00002060-200005000-00002. PMID 10821306
- [Background] Wang AY, Jaeger RJ, Yarkony GM, Turba RM. Cough in spinal cord injured patients: the relationship between motor level and peak expiratory flow. Spinal Cord. 1997 May;35(5):299-302. doi: 10.1038/sj.sc.3100370. PMID 9160454
- [Background] Schilero GJ, Radulovic M, Wecht JM, Spungen AM, Bauman WA, Lesser M. A center's experience: pulmonary function in spinal cord injury. Lung. 2014 Jun;192(3):339-46. doi: 10.1007/s00408-014-9575-8. Epub 2014 Apr 11. PMID 24723067
- [Background] Chamberlain JD, Meier S, Mader L, von Groote PM, Brinkhof MW. Mortality and longevity after a spinal cord injury: systematic review and meta-analysis. Neuroepidemiology. 2015;44(3):182-98. doi: 10.1159/000382079. Epub 2015 May 13. PMID 25997873
- [Background] Tollefsen E, Fondenes O. Respiratory complications associated with spinal cord injury. Tidsskr Nor Laegeforen. 2012 May 15;132(9):1111-4. doi: 10.4045/tidsskr.10.0922. English, Norwegian. PMID 22614314
- [Background] Liebscher T, Niedeggen A, Estel B, Seidl RO. Airway complications in traumatic lower cervical spinal cord injury: A retrospective study. J Spinal Cord Med. 2015 Sep;38(5):607-14. doi: 10.1179/2045772314Y.0000000254. Epub 2014 Aug 12. PMID 25117865
- [Background] Aarabi B, Harrop JS, Tator CH, Alexander M, Dettori JR, Grossman RG, Fehlings MG, Mirvis SE, Shanmuganathan K, Zacherl KM, Burau KD, Frankowski RF, Toups E, Shaffrey CI, Guest JD, Harkema SJ, Habashi NM, Andrews P, Johnson MM, Rosner MK. Predictors of pulmonary complications in blunt traumatic spinal cord injury. J Neurosurg Spine. 2012 Sep;17(1 Suppl):38-45. doi: 10.3171/2012.4.AOSPINE1295. PMID 22985369
- [Background] Croce MA, Fabian TC, Waddle-Smith L, Maxwell RA. Identification of early predictors for post-traumatic pneumonia. Am Surg. 2001 Feb;67(2):105-10. PMID 11243529
- [Background] Postma K, Bussmann JB, Haisma JA, van der Woude LH, Bergen MP, Stam HJ. Predicting respiratory infection one year after inpatient rehabilitation with pulmonary function measured at discharge in persons with spinal cord injury. J Rehabil Med. 2009 Sep;41(9):729-33. doi: 10.2340/16501977-0410. PMID 19774306
- [Background] Berlowitz DJ, Tamplin J. Respiratory muscle training for cervical spinal cord injury. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD008507. doi: 10.1002/14651858.CD008507.pub2. PMID 23881660
- [Background] Mueller G, Hopman MT, Perret C. Comparison of respiratory muscle training methods in individuals with motor and sensory complete tetraplegia: a randomized controlled trial. J Rehabil Med. 2013 Mar;45(3):248-53. doi: 10.2340/16501977-1097. PMID 23389554
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Derived] Raab AM, Brinkhof MWG, Berlowitz DJ, Postma K, Gobets D, Hirschfeld S, Hopman MTE, Huber B, Hund-Georgiadis M, Jordan X, Schubert M, Wildburger R, Mueller G. Respiratory function and respiratory complications in spinal cord injury: protocol for a prospective, multicentre cohort study in high-income countries. BMJ Open. 2020 Nov 5;10(11):e038204. doi: 10.1136/bmjopen-2020-038204. PMID 33154049

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants had to be excluded before start
Groups:
- Inpatient Rehab: all new SCI in inpatient rehabilitation
Period: Overall Study
Arm/Group | Inpatient Rehab
Started | 546
Completed | 503
Not Completed | 43

BASELINE CHARACTERISTICS:
Arm/Group | Inpatient Rehab
Number analyzed (Participants) | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 328
  >=65 years | 175
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 382
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 251
  Australia | 55
  Austria | 94
  Germany | 20
  Netherlands | 83

OUTCOME MEASURES:

1. Primary Outcome: Pneumonia
Description: occurrence of pneumonia
Time Frame: From date of spinal cord injury until discharge from primary rehabilitation (i.e. individual time window of observation from a few weeks to about 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Rehab
Number analyzed (Participants) | 503
Participants | 70

2. Secondary Outcome: Respiratory Function Measurements
Description: The various lung parameters thus include, vital capacity (FVC), forced expiratory volume in 1 second (FEV1), peak expiratory flow (PEF) and peak cough flow (PCF).
  The measurement of the lung function will be conducted in sitting position in the own wheelchair or for pedestrians on a chair and lasts at most 15 minutes.
  The peak cough flow (PCF) will be measured by having the person cough as forcefully as possible through a peak flow meter.
  The greatest value of each lung function parameter will be used for analysis.
Time Frame: measured at inclusion at 28±12 days post injury (time window) or at 84±14 days post injury (time window) - first measurement of each patient used for analysis
Population: all participants who had measurements
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- With Pneumonia: all study participants who experienced at least one pneumonia event during inpatient rehabilitation
- Without Pneumonia: all study participants without any pneumonia diagnosis during inpatient rehabilitation
Arm/Group | With Pneumonia | Without Pneumonia
Number analyzed (Participants) | 65 | 425
Liters
  FVC: number analyzed (Participants) | 65 | 423
  FVC | 2.60 (1.10) | 3.18 (1.09)
  FEV1: number analyzed (Participants) | 65 | 423
  FEV1 | 2.20 (0.90) | 2.59 (0.95)
  PEF: number analyzed (Participants) | 65 | 423
  PEF | 292.4 (130.1) | 359.3 (135.0)
  PCF: number analyzed (Participants) | 65 | 411
  PCF | 319.9 (150.0) | 374.5 (140.5)

3. Secondary Outcome: Mortality Due to Pneumonia
Description: Mortality will be defined as pneumonia-related, if a prevailing event of pneumonia was clinically resolved as the initiating factor of the cascade of morbid events leading directly to death. Similarly, other causes of death will be recorded as part of all-cause mortality and as potentially competing risks of death.
Time Frame: From date of spinal cord injury until discharge from inpatient rehabilitation (i.e. individual time window of observation from a few weeks to about 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | With Pneumonia | Without Pneumonia
Number analyzed (Participants) | 70 | 433
Participants | 1 | 1

4. Other Pre Specified Outcome: Quality of Life in General
Description: Quality of life (Qol) will be evaluated using the Quality of Life Basic Data Set of the International Spinal Cord Injury Datasets. This measurement instrument accepts (Qol) as a multi-facetted concept and includes three questions as to capture general quality of life (overall well-being), rating of physical health, and satisfaction with psychological health.
Time Frame: in days post injury: T1:28±12; T2:84±14, T3:150±18; T4:15 days before discharge until discharge
Reporting Status: Not Posted

5. Secondary Outcome: Respiratory Muscle Strength
Description: maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP)
  The measurement will be conducted in sitting position in the own wheelchair or for pedestrians on a chair . The measurements will be conducted with a device for respiratory pressure measurement in which the patient has to inhale and exhale through a mouthpiece. Each measurement of the inspiration and expiration will be repeated 3 times per measurement time.
  The greatest value of each parameter will be used for analysis.
Time Frame: as for outcome 2
Population: all participants who had measurements
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | With Pneumonia | Without Pneumonia
Number analyzed (Participants) | 65 | 425
cmH2O
  MIP | 60.4 (24.8) | 72.4 (29.4)
  MEP | 50.5 (24.8) | 78.0 (37.2)

ADVERSE EVENTS:
Time Frame: between start of T1 (28±12 days post injury) and end of T4 (up to 15 days before of discharge) (i.e. individual time window of observation from a few weeks to about 1 year)
Description: only serious adverse events were collected
Arm/Group | Inpatient Rehab
All-Cause Mortality (participants affected / at risk) | 2/503
Serious Adverse Events (participants affected / at risk) | 0/503
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT02891096/Prot_SAP_000.pdf